CLINICAL TRIAL: NCT03559842
Title: Sleeve-gastrectomy Efficacy in the Treatment of Metabolic and Vascular Dysfunction of Morbid Obese Patient With a Focus on the Role of Inflammation
Brief Title: Sleeve-gastrectomy Efficacy in Morbid Obese Patient With a Focus on the Role of Inflammation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Maria Anastasia Ricci, Principal Investigator, University Of Perugia
Other Study IDs: 2017-15
Record Dates: First submitted 2018-05-19; First posted 2018-06-18 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, serum, plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery patients: Obese patients undergoing laparoscopic sleeve gastrectomy
- Non-surgery patients: Obese patients not undergoing laparoscopic sleeve gastrectomy (delayed or refused proposed treatment)

SUMMARY:
Despite the wide range of studies concerning the positive effects of bariatric surgery on metabolic state of morbid obese patient, it is necessary to further investigate the specific role of the "sleeve-gastrectomy" intervention, going not only to research results in terms of safety or efficacy on the treatment of comorbidities, but also aimed to understand whether the improvement of metabolic and cardiovascular parameters is due to total weight loss or rather to visceral fat loss, and how much of this improvement is attributable to changes in inflammatory status. The primary endpoint of the study is to evaluate the effect of sleeve-gastrectomy on metabolic parameters (glyco-lipidic assessment, vitamins), bone-remodelling parameters (vitamin D, parathormone) and cardiovascular parameters (blood pressure, flow-mediated dilation, indexed left ventricular mass, inter-ventricular septum, carotid intima-media thickness) in a large obese population on the basis of total weight loss (TWL), variation of visceral fat area (VFA), variation of peri-renal fat thickness and insulin resistance index ("Homeostasis Model Assessment-insulin resistance" - HOMA). In addition the investigators set themselves the objective of assessing whether the presence of comorbidities (diabetes and hypertension) can influence the effects of the intervention on the above parameters, and whether the levels of the NETs and of adipokines such as chemerin in the pre- and post-intervention can correlate with the metabolic-vascular dysfunction, and play a role in its eventual improvement.

ELIGIBILITY:
Inclusion Criteria:

- BMI ≥ 40 kg / m2 (or ≥ 35 kg / m2 with at least one comorbidity), aged between 18 and 65 years.

Exclusion Criteria:

* renal or hepatic impairment
* heart failure (New York Heart Association - NYHA II-IV)
* secondary causes of obesity
* major psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Morbid obese patients with BMI ≥ 40 kg / m2 (or ≥ 35 kg / m2 with at least one comorbidity)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2017-05-04 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
flow-mediated dilation | One year
  ultrasound evaluation
obesity-related cardiomyopathy | One year
  cardiac ultrasonography
insulin resistance | One year
  HOMA index
ectopic adiposity | One year
  ultrasound evaluation of visceral fat
inflammation | One year
  high sensitivity C reactive protein, sclerostin, osteopontin, cathepsin K, IL-10
blood pressure | One year
  systolic and diastolic blood pressure
carotid intima-media thickness | One year
  ultrasound evaluation
microcirculatory function | One year
  Laser-Doppler flowmetry
aortic stiffness | One year
  tonometry
cardiovascular assessment | One year
  anti-hypertensive therapy variation (number of drugs)
dyslipidemia | One year
  total cholesterol, triglycerides, HDL, LDL
liver function | One year
  Evaluation of "Non-alcoholic fatty liver disease" (NAFLD) fibrosis score according to the following formula:
  -1.675 + 0.037 × age (years) + 0.094 × BMI (kg/m2) + 1.13 × IFG/diabetes (yes = 1, no = 0) + 0.99 × AST/ALT ratio - 0.013 × platelet (×109/l) - 0.66 × albumin (g/dl).
  Cutoffs:
  NAFLD Score < -1.455 = low grade fibrosis; NAFLD Score -1.455 - 0.675 = indeterminate score; NAFLD Score > 0.675 = high grade fibrosis.
biliary acid and sterols assessment | One year
  laboratory analysis
bone metabolism assessment | One year
  vitamin D, PTH
nutritional assessment | One year
  sideremia, vitamin B12, folates
adipose tissue quantification | One year
  bioimpedentiometry
adipokines | One year
  chemerin, leptin and adiponectin plasmatic dosage
NETs | One year
  "Neutrophil extracellular traps" dosage

SECONDARY OUTCOMES:
inflammatory bone remodeling markers | One year
  sclerostin, osteopontin, cathepsin K
macrophages commitment markers | One year
  interleukin-10

CONTACTS AND LOCATIONS:
Locations (1):
- Internal Medicine, Perugia, Italy